CLINICAL TRIAL: NCT07236996
Title: Evaluation of the Health Effects of the Air Purifier in Preterm Infants After Discharge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KMUHIRB-SV(I)-20210024
Record Dates: First submitted 2025-07-03; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-04

CONDITIONS: Premature - Weight 1000g-2499g or Gestation of 28-37weeks; Premature Birth
MeSH Terms: conditions — Premature Birth | interventions — Air Filters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comparison of Air Purifier Intervention and Frequency of Medical Visits (Experimental): Study Arm: Experimental (Air Purifier On) vs. No Intervention (Air Purifier Off）
  Interventions: Device: air purifier

INTERVENTIONS:
Device: air purifier — air purifier with mechanism of PCO plus three in one filters (Pre-filter/High-Efficiency Activated Carbon/High-Efficiency Particulate Air (HEPA) )

SUMMARY:
Participant's baby was born prematurely and had underdeveloped lungs at birth. Most premature infants require mechanical ventilation after birth, which increases the risk of lung injury and may lead to varying degrees of bronchopulmonary dysplasia (BPD). Investigators believe that introducing an air purifier into your home environment after Participant's baby is discharged could help improve their lung development.

This study aims to non-invasively measure baby's transcutaneous carbon dioxide (PtcCO₂) levels and blood oxygen saturation (SpO₂) at home, both with and without the use of an air purifier. In addition, investigators will collect data from Kaohsiung Medical University Hospital medical records regarding the number of visits, respiratory status, height, weight, head circumference, and developmental progress. Health questionnaires will also be administered to assess changes in health outcomes and provide recommendations on improving indoor air quality in Participant's home.

ELIGIBILITY:
Inclusion Criteria:Children aged 0 to 6 years who were born at less than 37 weeks of gestation.

-

Exclusion Criteria:Children born at more than 37 weeks of gestation.

-

Max Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in particulate matter concentrations (PM₁, PM₂.₅, PM₄, PM₁₀, TSP) | Baseline and up to 3 weeks after intervention
  Indoor concentrations of PM₁, PM₂.₅, PM₄, PM₁₀, and total suspended particles (TSP) will be measured before and after the use of an air purifier.
  Unit of Measure:µg/m³
Change in gaseous pollutant concentrations (CH₂O, NO₂, CO, SO₂, VOC, CO₂) | Baseline and up to 3 weeks after intervention
  Indoor gaseous pollutants, including formaldehyde (CH₂O), nitrogen dioxide (NO₂), carbon monoxide (CO), sulfur dioxide (SO₂), volatile organic compounds (VOC), and carbon dioxide (CO₂), will be measured before and after the intervention.
  Unit of Measure: ppm
Change in microbial concentrations (bacteria, fungi, Gram-positive, Gram-negative) | Baseline and up to 3 weeks after intervention
  Airborne microbial concentrations, including total bacteria, total fungi, Gram-positive bacteria, and Gram-negative bacteria, will be assessed before and after the use of an air purifier.
  Unit of Measure: CFU/m³
Change in lung function parameters (SVC, FVC, FEV₁,） | Baseline and up to 3 weeks after intervention
  Change in lung volumes including Slow Vital Capacity (SVC), Forced Vital Capacity (FVC), and Forced Expiratory Volume in 1 second (FEV₁) of household members living with preterm infants. Measurements will be taken before and after the intervention.
  Unit of Measure: Liters (L)
Change in Airflow Rates(MMEF,FEF25,FEF50,FEF75,PEF) | Baseline and up to 3 weeks after intervention
  Change in airflow parameters including Maximum Mid-Expiratory Flow (MMEF), Forced Expiratory Flow at 25% (FEF₂₅), 50% (FEF₅₀), and 75% (FEF₇₅) of FVC, and Peak Expiratory Flow (PEF) of household members living with preterm infants. Measurements will be taken before and after the intervention.
  Unit of Measure: Liters per second (L/s)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan